CLINICAL TRIAL: NCT01032772
Title: ChoicesPlus: Preconception Approach to Reducing Alcohol- and Tobacco-Exposed Pregnancy
Brief Title: ChoicesPlus: Reducing Alcohol- and Tobacco-Exposed Pregnancy
Acronym: ChoicesPlus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5U84DD000438 (NIH)
Record Dates: First submitted 2009-12-12; First posted 2009-12-15 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Alcohol Use; Smoking; Contraception
Keywords: alcohol-exposed pregnancy; tobacco-exposed pregnancy; alcohol; contraception; smoking; pregnancy
MeSH Terms: conditions — Alcohol Drinking; Smoking | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHOICES Plus Intervention (Experimental): A two session intervention utilizing a motivational interviewing approach to encourage changes in alcohol use, contraceptive use, and smoking. The interventions will (a) provide norms-based-but personalized-feedback, (b) encourage attendance at a contraceptive counseling visit, (c) encourage participation in the smoking cessation program, (c) increase motivation to change each of the target behaviors, (d) decrease temptation to engage in risk behaviors, (e) increase confidence to avoid risk behaviors, and (f) develop a personalized, tailored change plan.
  Interventions: Behavioral: Choices Plus
- Information (Active Comparator): Women in the information condition receive advice and educational material from the research assistant about women's health and related referrals.
  Interventions: Behavioral: Information

INTERVENTIONS:
Behavioral: Choices Plus — Participants in this condition will receive two brief, motivational-interviewing-based counseling sessions.
  Arms: CHOICES Plus Intervention
Behavioral: Information — Participants are provided with informational materials about healthy lifestyle and local resources.
  Other Names: Treatment As Usual
  Arms: Information

SUMMARY:
Choices Plus, a randomized controlled study, will determine the efficacy of the Project CHOICES intervention plus a referral to an evidence-based smoking cessation program in reducing the risk of alcohol- and tobacco-exposed pregnancies.

DETAILED DESCRIPTION:
This randomized controlled study will examine the effect of the ChoicesPlus intervention compared to Treatment as Usual (TAU) in: reducing alcohol use below established risk levels; increasing consistent use of effective contraception; increasing engagement in smoking cessation treatment and increasing smoking cessation. In addition, our examination of the incremental costs of the ChoicesPlus intervention (e.g., staff time, materials, administrative services, total medical charges pre- and post-intervention) will provide a basis for future cost/benefit analyses that will inform policymakers and healthcare organizations of the potential benefits of implementing ChoicesPlus. Results from this study will inform and advance future efforts in the service of promoting healthy prenatal behavior and reducing the prevalence of alcohol and tobacco-exposed pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Have no condition causing infertility
* Are not pregnant or planning to become pregnant in the next 9 months
* Have had vaginal intercourse during the previous 3 months with a fertile man without using effective contraception
* Are drinking at risk levels; and 5) are available for the follow-up period.

Exclusion Criteria:

* Infertile
* Pregnant
* Insufficient locator information
* Language other than English or Spanish

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 261 (Actual)
Dates: Start 2010-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Risk of alcohol-exposed pregnancy | 9 months
  Timeline Followback

SECONDARY OUTCOMES:
Marin Acculturation Scale, AUDIT, Time-Line Follow Back, University of Rhode Island Change Assessment Scale, Decisional Balance, Process of Change, Temptation, Confidence, Smoking Staging Algorithm, and Brief Symptom Inventory-18 | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary M Velasquez, Ph.D., Principal Investigator — University of Texas at Austin; Kirk von Sternberg, Ph.D., Principal Investigator — University of Texas at Austin
Locations (2):
- United States (2):
  - Settegast Health Center, Houston, Texas
  - Strawberry Health Center, Pasadena, Texas

REFERENCES:
- [Derived] Northrup TF, Stotts AL, Fischer SM, von Sternberg KL, Velasquez MM. Increased risk for alcohol- and other substance-exposed pregnancies among women who smoke tobacco: A secondary analysis of a primary care-based intervention. Tob Induc Dis. 2024 Jul 26;22. doi: 10.18332/tid/191107. eCollection 2024. PMID 39072280
- [Derived] Velasquez MM, von Sternberg KL, Floyd RL, Parrish D, Kowalchuk A, Stephens NS, Ostermeyer B, Green C, Seale JP, Mullen PD. Preventing Alcohol and Tobacco Exposed Pregnancies: CHOICES Plus in Primary Care. Am J Prev Med. 2017 Jul;53(1):85-95. doi: 10.1016/j.amepre.2017.02.012. Epub 2017 Apr 17. PMID 28427955